CLINICAL TRIAL: NCT00662623
Title: Enabling Sleep Apnea Patient-Centered Care Via an Internet Intervention
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Responsible Party: Principal Investigator, Carl J. Stepnowsky, Study PI, Veterans Medical Research Foundation
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS-17246-01
Record Dates: First submitted 2008-04-16; First posted 2008-04-21 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Sleep Apnea Syndromes
Keywords: Chronic Obstructive Sleep Apnea; Sleep Apnea; Sleep Apnea Treatment
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: i-PAP
- 2 (Active Comparator): Usual Care (Standard Care)
  Interventions: Behavioral: Usual Care (Standard Care)

INTERVENTIONS:
Behavioral: i-PAP — Internet Intervention based on wireless telemonitoring of CPAP data and patient-centered, collaborative care
  Arms: 1
Behavioral: Usual Care (Standard Care) — Pre-determined clinic visits and telephone support
  Arms: 2

SUMMARY:
The purpose of this study is to examine the effect of different methods of providing education about sleep apnea and continuous positive airway pressure therapy (CPAP) use and how that education might help to improve health outcomes and the amount of time CPAP is used.

DETAILED DESCRIPTION:
Poor treatment adherence with CPAP therapy is well-documented. Set against a backdrop of telemedicine applications that have grown as fast in unsubstantiated claims and assumptions of patient satisfaction, diagnostic accuracy, clinical efficacy, and cost-effectiveness as they have in technological sophistication and capabilities, the evaluative aspect of this proposal is designed as as a randomized, controlled clinical trial-Usual Care patients (control) versus i-PAP patients (intervention). An important empirical-methodological advantage of the project is the objective measurement of CPAP adherence, which is measured by internal microprocessor as the "amount of time CPAP is used at the prescribed pressure." This objective measurement allows feedback of treatment adherence and efficacy to both patient and provider, and the i-PAP intervention was designed around this central feature.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* confirmed diagnosis of OSA
* being newly prescribed CPAP therapy
* having chronic symptoms as noted on screening symptom checklist
* fluency in English

Exclusion Criteria:

* cognitive impairment sufficient to cause inability to complete the protocol (MMSE < 24/30)
* residence in a geographical area outside of San Diego County
* fatal comorbidity (life expectancy less than 6 months as indicated by treating physician)
* significant documented substance/chemical abuse or other participant circumstances that, in the opinion of a consensus of study team, would interfere with the safety of a prospective participant or their need for treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
CPAP Adherence | 4 months

SECONDARY OUTCOMES:
Quality of patient-centered collaborative care | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Carl J. Stepnowsky, PhD, Principal Investigator — Veterans Medical Research Foundation
Locations (1):
- Veterans Medical Research Foundation, San Diego, California, United States